CLINICAL TRIAL: NCT03003754
Title: Supervised Exercise-training in Children With Insulin Resistance or Healthy Metabolic Profile: Cardiometabolic Risk Factors and Muscular Strength Changes in Responders and Non Responders
Brief Title: Supervised Exercise-training in Children With Insulin Resistance or Healthy Metabolic Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas (Other)
Collaborators: Healthcare Center Tomas Rojas (Other); Health Service of Los Ríos by the Health promotion program (Unknown); Universidad Pública de Navarra (Other); Universidad del Rosario (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-12-22
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Metabolism Disorder; Insulin Sensitivity; Obesity, Pediatric
MeSH Terms: conditions — Metabolic Diseases; Insulin Resistance; Pediatric Obesity | interventions — Resistance Training; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Intensity Training (HIT) + Resistance Training (RT) (Experimental): To HIT program will be use cycle ergometers adapted for children (OXFORDTM, model BE2601, OXOFORD Inc, Santiago, Chile) were used. Each participant performed a range of 8 to 14 cycling intervals during the intervention period. The time of each work interval cycling will be increased progressively weekly, and ranged between 40-60 s (40 s weeks 1-2; 50 s weeks 3-5; 60 s week 6), with 120 s of passive rest (over the bicycle without movement) between each interval of work.
  The RT will consist in voluntary concentric/eccentric exercise during 1 minute until to get a high subjective effort perception (i.e., between 8-10 points based on the modified and subjective Borg scale of 1 to 10 points. Subjects will perform 4 exercises (biceps curl, leg-extension, shoulders press, and upper row exercise) during 6-weeks.
  Interventions: Behavioral: High Intensity Training (HIT) + Resistance Training (RT)
- Control group (Active Comparator): We will compare within each group (G)-1, G-2, and G-3 sub-group according to both RT and HIT intervention both pre-post changes as well as if are there some anthropometric, cardiovascular, and performance variable predicting changes in homeostasis model assessment (HOMA-IR).
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: High Intensity Training (HIT) + Resistance Training (RT) — Exercise will be performed at three sessions per week. Post statistical analyses will be including analyses by the 3 sub-groups proposed. All sessions will be supervised by an exercise physiologist during 6 weeks.
  Arms: High Intensity Training (HIT) + Resistance Training (RT)
Behavioral: Control group — Post statistical analyses will be including analyses by the 3 sub-groups proposed Exercise will be performed at three sessions per week. All sessions will be supervised by an exercise physiologist during 6 weeks.
  Arms: Control group

SUMMARY:
Despite exercise training decrease blood fasting glycemia in 'average' terms, there is a wide interindividual variability after exercise training explored mainly in adults but not in children. Thus, is yet unknown what baseline health status as well as the influence of what health variable may produce more/less non-responder (NR) prevalence (i.e., percentage of subjects who experienced a non-change/worsened response after training in some metabolic outcomes) after exercise training in school children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of insulin resistance by one of three plasmatic glucose control: HOMA-IR ≥3.0,
* Fasting insulin levels ≥15 µUI/dL or fasting glucose ≥100 and ≤126 mg/dL within the enrolment stage applied at school (i.e., ≤3 months),
* Physical inactivity (volume of ≤60 min/day of moderate physical activity),
* To be participating of regular practical physical education classes at school (i.e., 90 min/week),
* Living only in urban areas.

Exclusion Criteria:

* Potential medical, musculoskeletal problems or a familial history of T2DM,
* Ischemic disease,
* Arrhythmia,
* Asthma,
* Utilization of drugs that modulate the metabolic and respiratory control.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in plasma homeostasis model assessment (HOMA-IR) | Baseline and 6 weeks immediately after the interventions ends

SECONDARY OUTCOMES:
Change from Baseline in body mass | Baseline and 6 weeks immediately after the interventions ends
Change from Baseline in body mass index | Baseline and 6 weeks immediately after the interventions ends
Change from Baseline in waist circumference | Baseline and 6 weeks immediately after the interventions ends
Change from Baseline in fat mass | Baseline and 6 weeks immediately after the interventions ends
Change from Baseline in blood pressure | Baseline and 6 weeks immediately after the interventions ends
Change from Baseline in fasting glucose | Baseline and 6 weeks immediately after the interventions ends
Change from Baseline in fasting insulin | Baseline and 6 weeks immediately after the interventions ends
Change from Baseline in one maximum repetition strength test of leg-extension exercise | Baseline and 6 weeks immediately after the interventions ends
Change from Baseline in one maximum repetition strength test of shoulder press exercise | Baseline and 6 weeks immediately after the interventions ends
Change from Baseline in one maximum repetition strength test of upper-row exercise | Baseline and 6 weeks immediately after the interventions ends
Change from Baseline in one maximum repetition strength test of biceps curl exercise | Baseline and 6 weeks immediately after the interventions ends

CONTACTS AND LOCATIONS:
Locations (1):
- Robinson Ramírez-Vélez, Bogota Distrito Especial, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarez C, Ramirez-Campillo R, Ramirez-Velez R, Martinez C, Castro-Sepulveda M, Alonso-Martinez A, Izquierdo M. Metabolic effects of resistance or high-intensity interval training among glycemic control-nonresponsive children with insulin resistance. Int J Obes (Lond). 2018 Jan;42(1):79-87. doi: 10.1038/ijo.2017.177. Epub 2017 Jul 31. PMID 28757639